CLINICAL TRIAL: NCT04871724
Title: A Non-Randomized, Open-Label, Drug-Drug Interaction Study to Evaluate the Effects of Fluconazole on the Pharmacokinetics and Safety of EDP-938 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study Between Fluconazole and EDP-938 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDP 938-007
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: RSV Infection
Keywords: drug-drug interaction
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EDP-938 and Fluconazole interaction (Experimental)
  Interventions: Drug: EDP-938; Drug: Fluconazole

INTERVENTIONS:
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Days 1 and 14
Drug: Fluconazole — Subjects will receive fluconazole once daily on Days 5 to 18

SUMMARY:
A Non-Randomized, Open-Label, Drug-Drug Interaction Study to Evaluate the Effects of Fluconazole on the Pharmacokinetics and Safety of EDP-938 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP 938.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at Screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.
* Clinically significant history of drug sensitivity or allergy to fluconazole or other azole antifungals

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-938 with and without coadministration with fluconazole | Up to 19 days
AUC of EDP-938 with and without coadministration with fluconazole | Up to 19 days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 25 Days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No